CLINICAL TRIAL: NCT00239603
Title: Clinical Investigation of the OV-Watch™ Personal Fertility Monitor for Women Undergoing Ovulation Induction With Clomiphene Citrate.
Brief Title: Efficacy Study of the OV-Watch™ Personal Fertility Monitor for Women Using Clomiphene Citrate.
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: HealthWatchSystems, Inc. (Industry)
Other Study IDs: 867-2005
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2007-04-17 (Estimated); Status verified 2007-04

CONDITIONS: Infertility; Anovulation; Polycystic Ovary Syndrome
Keywords: OV-Watch; fertility monitor; ovulation induction; clomiphene citrate; anovulation; infertility
MeSH Terms: conditions — Infertility; Anovulation; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: OV-Watch

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the OV-Watch to predict ovulation while women are taking clomiphene citrate.

DETAILED DESCRIPTION:
At any given time, there are 10-15% of American couples with infertility. A problem with ovulation (releasing an egg) is one of the most common causes of female infertility. The frequency and timing of intercourse is important because the best chance of pregnancy occurs around the time of ovulation. The days that pregnancy is most likely to occur with intercourse is referred to as the "fertile window".

The fertile window lasts for 6 days. It starts 4 days before ovulation and continues through the day after ovulation. Intercourse on the day of ovulation gives the highest chance of getting pregnant. However, intercourse up to 4 days before ovulation can still result in pregnancy because sperm can survive for up to 6 days in the reproductive tract of a woman.

Urinary testing for the luteinizing hormone (LH) surge is the most common method for predicting ovulation. The LH surge precedes ovulation by about 36 hours. When LH is detected, this gives a couple only 2 days to have intercourse that may result in fertilization.

The OV-Watch is an FDA approved device that has been shown to predict ovulation 5 days in advance for women who ovulate regularly. This wristwatch-like device is worn daily to detects changes in sweat ions. The device allows for earlier detection of the fertile window, giving the couple more opportunities to conceive.

For women who do not ovulate on their own or ovulate irregularly, medication can be taken to help make eggs and ovulate. Clomiphene citrate is the most commonly used medication for this. We plan to study the effectiveness of the OV-Watch in women who are undergoing ovulation induction with clomiphene citrate and will compare the results to standard urinary LH testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to participate must be between the age of 21 and 42.
* Patient must demonstrate ability to follow standard clomiphene citrate ovulation induction protocol and wear the OV-Watch™ correctly.
* Intact uterus and at least one ovary must be present.
* Patients must be diagnosed with anovulation (lack of ovulation) that is not caused by hypothalamic amenorrhea or premature ovarian failure.
* A hysterosalpingogram must be performed to demonstrate at least one patent fallopian tube. The uterine cavity must also appear normal on this study.
* The male partner or sperm donor must demonstrate an acceptable concentration and motility of sperm.

Exclusion Criteria:

* 12 or more previous treatment cycles using clomiphene citrate.
* Any condition where the use of clomiphene is contraindicated, such as breast cancer or liver disease.
* Any other hormonal disease that may be secondarily causing anovulation, such as thyroid disorder or hyperprolactinemia.
* Amenorrhea caused by premature ovarian failure or hypothalamic amenorrhea.
* Any active genital tract infection will need to be treated with antibiotics before undergoing ovulation induction.

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-10; Study Completion 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Celia E Dominguez, MD, Principal Investigator — Emory Reproductive Center
Locations (1):
- Emory Reproductive Center, Crawford Long Hospital, Atlanta, Georgia, United States